CLINICAL TRIAL: NCT05431920
Title: Effects of Vitamin D3 Supplementation in Asthma Control, Pulmonary Function and Th17 Inflammatory Biomarkers in Adolescents With Asthma, Obesity and Vitamin D Deficiency: a Randomized Clinical Trial
Brief Title: Effects of Vitamin D Supplementation in Adolescents With Asthma, Obesity and Vitamin D Deficiency.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Blanca Estela Del Rio Navarro, Alternate investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIM/2021/023
Record Dates: First submitted 2022-06-08; First posted 2022-06-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Non-allergic Asthma; Obesity; Vitamin D Deficiency
Keywords: asthma; obesity; non allergic asthma; adolescents; vitamin D; 25-hydroxyvitamin D
MeSH Terms: conditions — Obesity; Vitamin D Deficiency; Asthma | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Adolescents with non-allergic asthma, obesity and insufficiency/deficiency of vitamin D will be randomized in block (33 groups with 8 patients), 2 arms of 132 patients each: the experimental group will receive a single dose of 50,000 IU followed by 4,000 IU daily of vitamin D for three months, and the control group will receive 2,000 IU daily of vitamin D for three months.
  Each patient will have a monthly follow up (weeks 4, 8 and 12 after the beginning of the intervention) with physical examination, questionnaire to evaluate asthma control, asthma control test and pediatric asthma quality of life questionnaire (PAQLQ), a spirometry with bronchodilator, 10 ml of peripheral blood to measure plasmatic concentration of 25-hydroxyvitamin D with electrochemiluminescence, Th17 inflammatory biomarkers and allergy skin tests (at the beginning and end of the intervention) and each visit will be a capsule count and a registration of adverse effects.
Who Masked: Care Provider
Masking Description: The masking will be done by a care provider. Each patient will have a randomly assigned envelope with the corresponding vitamin D dose, defining the allocated arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Vitamin D3: single 50,000 IU loading dose + 4,000 IU daily dose for three months
  Interventions: Dietary Supplement: Vitamin D₃ (25-hydroxy vitamin D)
- Active control (Active Comparator): Vitamin D3: 2,000 IU daily dose for three months
  Interventions: Dietary Supplement: Vitamin D₃ (25-hydroxy vitamin D)

INTERVENTIONS:
Dietary Supplement: Vitamin D₃ (25-hydroxy vitamin D) — Vitamin D3 oral supplementation
  Arms: Experimental
Dietary Supplement: Vitamin D₃ (25-hydroxy vitamin D) — Vitamin D3 oral supplementation
  Arms: Active control

SUMMARY:
Obesity has been associated with a specific non-allergic asthma phenotype and to a deficiency of vitamin D in at least 90% of the pediatric population. Adolescents with non-allergic asthma and vitamin D deficiency have up to six times the risk [OR: 6.2 (IC95% 2.0-21.6), p=0.002] of having a severe asthmatic crisis and do not respond adequately to inhaled steroid treatment.

To evaluate the effect of oral vitamin D3 supplementation with 50,000 IU single dose and 4,000 IU daily vs 2,000 IU daily on the Asthma Control Questionnaire score, number and incidence of asthmatic crisis, lung function, and Th17 inflammatory biomarkers in adolescents with asthma associated to obesity and vitamin D insufficiency/deficiency for three months.

DETAILED DESCRIPTION:
Randomized controlled, double-blind, parallel (2 arms), clinical trial. Eligibility criteria: adolescents (12-17 years old), with obesity, vitamin D deficiency (<30 ng/dl), controlled or partially controlled or uncontrolled asthma according to GINA 2020 criteria and confirmed with a spirometry, with negative allergy skin test.

To each patient it will be performed a medical history, physical examination, asthma control questionnaire, a spirometry (with bronchodilator), as well as a peripheral blood sample collection of 10 ml to measure Th17 inflammatory biomarkers by chemiluminescence immunoassay and quantitative polymerase chain reaction (genetic expression of 18 cytokines) and 25-hydroxyvitamin D plasmatic concentration with electrochemiluminescence.

Patients will be randomized by block and assigned to one of two intervention arms. Each intervention arm will have a total sample of 132 patients. Experimental group will receive a single dose of 50,000 IU and 4,000 IU of vitamin D daily for 3 months. On the other hand, the active control group will receive 2,000 IU daily for 3 months. Patients will be followed up and cited every month for clinical assessment, asthma control (ACQ) questionnaire application, spirometry (with bronchodilator) and peripheral blood sample collection to determine the plasma concentration of 25-hydroxyvitamin D and Th17 inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of 12 to 17 years old.
* Diagnosis of exogen obesity with a body mass index (BMI) greater than percentile 95 for age and sex, according to the Center for Disease Control and Prevention (CDC) graphics, that precedes the diagnosis of asthma.
* Plasmatic concentration of 25-hydroxyvitamin D less than 30 ng/ml at screening visit based on local laboratory test.
* Physician-diagnosed asthma, with more than 6 months of evolution, based on medical history, physical examination, clinical criteria according to the Global Initiative For Asthma 2020 (GINA) and confirmed with a spirometry with reversibility after the administration of a bronchodilator.
* Asthma severity (intermittent or mild persistent or moderate persistent) according to the National Asthma Education and Prevention Program (NAEPP) and classified as controlled, partly controlled or uncontrolled according to GINA 2020.
* Negative allergic skin tests.

Exclusion Criteria:

* History of systemic or chronic degenerative disease (renal, pulmonar, cardiovascular, infectious, muscular, immunological, hypertension, diabetes mellitus, cancer, nonalcoholic fatty liver disease).
* Current treatment with immunomodulators or immunostimulants, up to 6 months before the intervention.
* History of adverse effects to vitamin D.
* Treatment with oral steroids 3 months previous to the enrollment.
* Active smoking.

Elimination criteria:

* Parents, tutors, legal guardians or participants that decide to withdraw from the study any time.
* Pregnancy during study.
* Severe adverse effects to vitamin D.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of vitamin D supplementation daily for three months on asthma symptoms. | 12 weeks
  Evaluate the effects of vitamin D supplementation, with a single dose of 50,000 IU and 4,000 IU daily for three months, on asthma symptoms improvement (reduction of 0.5 in score compared to baseline), assessed by an asthma control questionnaire [score range from 0 (fully controlled) to 6 (severely uncontrolled)], compared to a dose of 2,000 IU daily.

SECONDARY OUTCOMES:
Evaluate the effects of vitamin D supplementation daily for three months on the incidence of asthmatic crisis. | 12 weeks
  Evaluate the effects of vitamin D supplementation, with a single dose 50,000 IU and 4,000 IU daily for three months, on asthma symptoms evaluated the incidence of asthmatic crisis compared to a dose of 2,000 IU daily.

OTHER OUTCOMES:
Evaluate the effects of vitamin D supplementation daily for three months on lung function. | 12 weeks
  Evaluate the effects of vitamin D supplementation, with a single dose 50,000 IU and 4,000 IU daily for three months, on lung function (Forced expiratory volume in the first second, 5% volume increase compared to baseline) compared to a dose of 2,000 IU daily.
Evaluate the effects of vitamin D supplementation for three months on IL-17A inflammatory biomarker. | 12 weeks
  Evaluate the effects of vitamin D supplementation, with a single dose of 50,000 IU and 4,000 IU daily for three months, on IL-17A (decrease of 5 pg/ml) compared to a dose of 2,000 IU daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil de México Federico Gómez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No